CLINICAL TRIAL: NCT00585559
Title: Inhibition of Lipid Peroxidation and Cerebral Vasospasm by an Acetaminophen-Based Regimen in Patients With Aneurysmal Subarachnoid Hemorrhage
Brief Title: Acetaminophen in aSAH to Inhibit Lipid Peroxidation and Cerebral Vasospasm
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Matthew Fusco, Assistant Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIH P50 GM015431; VUMCIRB060556; P50GM015431 (NIH)
Record Dates: First submitted 2007-12-26; First posted 2008-01-03 (Estimated); Results first posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-03

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage; Cerebral Vasospasm
Keywords: Lipid; Peroxidation; N-Acetylcysteine; Acetaminophen; Vasospasm
MeSH Terms: conditions — Subarachnoid Hemorrhage; Vasospasm, Intracranial | interventions — Acetaminophen; Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Placebos for acetaminophen and N-acetylcysteine (Placebo Comparator): Placebos for acetaminophen and N-acetylcysteine
  Interventions: Drug: Placebos for acetaminophen and N-acetylcysteine
- Acetaminophen and N-acetylcysteine placebo (Active Comparator): Acetaminophen 1 gm every 6 hours and N-acetylcysteine placebo
  Interventions: Drug: APAP 1 gm every 6 hours and N-acetylcysteine placebo
- N-acetylcysteine and acetaminophen (Active Comparator): N-acetylcysteine IV infusion at 0.5 gm hourly and acetaminophen placebo
  Interventions: Drug: NAC IV infusion at 0.5 gm hourly and APAP placebo
- Acetaminophen 1 Gram and N-acetylcysteine (Active Comparator): Acetaminophen 1 gm every 6 hours, plus N-acetylcysteine IV infusion at 0.5 gm hourly
  Interventions: Drug: APAP 1 gm q6 hours, plus NAC IV infusion at 0.5 gm hourly
- Acetaminophen 1.5 Gram and N-acetylcysteine (Active Comparator): Acetaminophen 1.5 gm every 6 hours, plus N-acetylcysteine IV infusion at 0.5 gm hourly
  Interventions: Drug: APAP 1.5 gm q6 hours, plus NAC IV infusion at 0.5 gm hourly

INTERVENTIONS:
Drug: Placebos for acetaminophen and N-acetylcysteine — Placebos for acetaminophen and N-acetylcysteine
  Arms: Placebos for acetaminophen and N-acetylcysteine
Drug: APAP 1 gm every 6 hours and N-acetylcysteine placebo — Acetaminophen 1 gm every 6 hours and N-acetylcysteine placebo
  Arms: Acetaminophen and N-acetylcysteine placebo
Drug: NAC IV infusion at 0.5 gm hourly and APAP placebo — N-acetylcysteine IV infusion at 0.5 gm hourly and acetaminophen placebo
  Arms: N-acetylcysteine and acetaminophen
Drug: APAP 1 gm q6 hours, plus NAC IV infusion at 0.5 gm hourly — Acetaminophen 1 gm every 6 hours, plus N-acetylcysteine IV infusion at 0.5 gm hourly
  Arms: Acetaminophen 1 Gram and N-acetylcysteine
Drug: APAP 1.5 gm q6 hours, plus NAC IV infusion at 0.5 gm hourly — Acetaminophen 1.5 gm every 6 hours, plus N-acetylcysteine IV infusion at 0.5 gm hourly
  Arms: Acetaminophen 1.5 Gram and N-acetylcysteine

SUMMARY:
The objective of this study is to determine whether acetaminophen (APAP), N-acetylcysteine (NAC), and APAP in combination with NAC will inhibit lipid peroxidation in aneurysmal subarachnoid hemorrhage (aSAH), utilizing F2-IsoPs as biomarkers for lipid peroxidation.

DETAILED DESCRIPTION:
Aneurysmal subarachnoid hemorrhage (aSAH) is an often devastating form of stroke with high morbidity and mortality despite advances in surgical management. Approximately 30,000 patients annually suffer aSAH in the U.S. For patients who survive the initial subarachnoid hemorrhage, delayed cerebral vasospasm occurring from days 4-14 is the greatest cause of neurological disability and death. A growing body of evidence incriminates hemoprotein-catalyzed lipid peroxidation as the mediator of the vasospasm.

Hemoglobin released from lysed red cells in the subarachnoid space becomes oxidized, in which state it acts as a pseudoperoxidase and generates the protein radicals that induce lipid peroxidation. F2-isoprostanes formed by this lipid peroxidation are highly potent constrictors of cerebral arterioles. We have demonstrated a more than 5 fold mean increase in F2-isoprostanes in the cerebrospinal fluid of patients with aSAH; this increase is maximal at the time of delayed vasospasm, and the level of increase is a function of the severity of the aSAH. We hypothesize that such vasoconstrictors are major contributors to the vasospasm produced by the hemoproteins, hemoglobin and myoglobin, in diseases in which they are released from their cellular confines.

We have discovered that acetaminophen (APAP) is a potent inhibitor of hemoprotein-catalyzed lipid peroxidation with an IC50 for hemoglobin of 15 uM, which is in the range of plasma levels resulting from therapeutic doses of the drug in humans. Acetaminophen acts by reducing the ferryl-oxo radical form of the heme, and thereby prevents formation of the hemoprotein radical that initiates lipid peroxidation. To assess proof of concept in vivo, we determined the effect of acetaminophen in a rat model of rhabdomyolysis in which renal failure results from intense vasospasm. Acetaminophen blocked lipid peroxidation in this model, and prevented the renal failure with a dose that produced plasma levels in the therapeutic range for humans.

We also have demonstrated that N-acetylcysteine (NAC) will inhibit hemoprotein-catalyzed lipid peroxidation. Moreover, NAC administration increases the levels of glutathione in vivo, and glutathione is a co-substrate for the glutathione peroxidases that can reduce the levels of peroxides in the environment of the aSAH . This is important as acetaminophen is most potent in inhibiting hemoprotein-catalyzed lipid peroxidation when peroxide concentrations are low. This concerted evidence is the basis for a hypothesis that NAC will augment the efficacy of acetaminophen as an inhibitor of hemoprotein-catalyzed lipid peroxidation in aSAH.

These finding provide the rationale for a pilot study seeking proof of the concept that acetaminophen-based regimens can inhibit lipid peroxidation in patients with subarachnoid hemorrhage. Lipid peroxidation will be determined by analysis of F2-isoprostanes in cerebrospinal fluid. If such inhibition is seen, that then would provide a basis for a larger multi-center investigation to assess the effect on clinical endpoints.

This pilot study will determine whether APAP, NAC, and APAP in combination with NAC will inhibit lipid peroxidation in aneurysmal subarachnoid hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

* Ages ≥ 20
* Fisher Grade III or III + IV SAH based upon admitting CT scan
* Aneurysm secured by either clipping or coiling within 72 hours of SAH
* Intracranial aneurysm confirmed by angiography or CTA
* Presence of ventriculostomy for external ventricular drainage (EVD) prior to randomization

Exclusion Criteria:

* Consent unobtainable
* Enrollment in another interventional study
* Patient is pregnant or lactating
* Known co-morbidities that could affect outcome of this study
* Contraindication to CTA
* Serum creatinine > 1.4
* Documented allergy to iodinated contrast that cannot be adequately treated with premedication
* Documented allergy and/or intolerance to ApAP
* Baseline liver disease
* History of recent alcohol abuse with documented ALT or AST above normal laboratory values
* Documented history of both malnutrition and decreased serum albumin below normal lab values
* Documented abnormal platelet count below normal lab values
* Documented abnormal PT or PTT above normal lab values
* History or evidence of active asthma
* Documented allergy and/or intolerance to N-acetylcysteine
* Currently taking phenytoin, carbamazepine, or phenobarbital
* Currently taking isoniazid (INH, Lanzid, Nydrazid)
* Severe life-threatening complications resulting from standard aneurysm treatments that will likely prevent completion of the study
* Patient unsuitable for the study, in the opinion of the investigator(s)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2007-04; Primary Completion 2023-10-26 (Actual); Study Completion 2023-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Fusco, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- N-acetylcysteine IV Infusion at 0.5 gm Hourly: N-acetylcysteine IV infusion at 0.5 gm hourly
- Placebo for N-acetylcysteine IV Infusion at 0.5 gm Hourly: Placebo for N-acetylcysteine IV infusion at 0.5 gm hourly
- Acetaminophen Plus N-acetylcysteine Infusion: Acetaminophen 1.5gm every 6 hours, plus N-acetylcysteine IV infusion at 0.5 gm hourly
Period: Overall Study
Arm/Group | N-acetylcysteine IV Infusion at 0.5 gm Hourly | Placebo for N-acetylcysteine IV Infusion at 0.5 gm Hourly | Acetaminophen Plus N-acetylcysteine Infusion
Started | 16 | 17 | 11
Completed | 16 | 17 | 11
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Aacetaminophen and N-acetylcysteine Infusion: Acetaminophen 1.5gm every 6 hours, plus N-acetylcysteine IV infusion at 0.5 gm hourly
- Total: Total of all reporting groups
Arm/Group | N-acetylcysteine IV Infusion at 0.5 gm Hourly | Placebo for N-acetylcysteine IV Infusion at 0.5 gm Hourly | Aacetaminophen and N-acetylcysteine Infusion | Total
Number analyzed (Participants) | 16 | 17 | 11 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 3 | 6
  >=65 years | 15 | 15 | 8 | 38
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 8 | 33
  Male | 4 | 4 | 3 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 2
  Not Hispanic or Latino | 16 | 16 | 10 | 42
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 1 | 5
  White | 15 | 13 | 9 | 37
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 16 | 17 | 11 | 44

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Vasospasm Based on Magnetic Resonance Angiography (MRA)
Description: Presence of vasospasm measured Magnetic Resonance Angiography (MRA). MRA measures the degree of arterial narrowing, with a higher score indicating more severe vasospasm. An MRA score of 84% sensitivity and 72% specificity is indicative of vasospasm.
Time Frame: 8 Days post subarachnoid hemorrhage (SAH) event
Population: No data for the prespecified outcome was analyzed due to the NIH-approved SAP that is powered for 34 placebo subjects and 34 N-acetylcysteine subjects to be able to reject the null hypothesis that the failure rates for placebo and N-acetylcysteine subjects are equal with probability (power) 0.8. Only 44 participants were randomized. As such, no data analysis will be completed for this underpowered study.
Groups:
- Acetaminophen Plus N-acetylcysteine IV Infusion: Acetaminophen 1.5gm every 6 hours, plus N-acetylcysteine IV infusion at 0.5 gm hourly
Arm/Group | N-acetylcysteine IV Infusion at 0.5 gm Hourly | Placebo for N-acetylcysteine IV Infusion at 0.5 gm Hourly | Acetaminophen Plus N-acetylcysteine IV Infusion
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: Number of Patients With Vasospasm Based on Computed Tomographic Angiography (CTA)
Description: Presence of vasospasm measured by Computed Tomographic Angiography (CTA). CTA scores range from 0 (no vasospasm) to 34, where a score of 10 or more is indicative of vasospasm.
Time Frame: 8 Days post subarachnoid hemorrhage (SAH) event
Population: as for outcome 1
Arm/Group | N-acetylcysteine IV Infusion at 0.5 gm Hourly | Placebo for N-acetylcysteine IV Infusion at 0.5 gm Hourly | Acetaminophen Plus N-acetylcysteine IV Infusion
Number analyzed (Participants) | 0 | 0 | 0

3. Primary Outcome: National Institutes of Health Stroke Scale (NIHSS) Score
Description: The scale measures the severity of symptoms associated with patient's stroke. It assesses the severity of impairments related to stroke. The impairments are graded on a 3-4 point scale with scores that range from 0-42. Patients with a higher score have a more severe impairment, and patients with a lower score have a less severe impairment.
Time Frame: 8 Days post subarachnoid hemorrhage (SAH) event
Population: as for outcome 1
Arm/Group | N-acetylcysteine IV Infusion at 0.5 gm Hourly | Placebo for N-acetylcysteine IV Infusion at 0.5 gm Hourly | Acetaminophen Plus N-acetylcysteine IV Infusion
Number analyzed (Participants) | 0 | 0 | 0

4. Primary Outcome: Modified Rankin Scale (MRS) Score
Description: The modified Rankin Scale (mRS) is used for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. The 7 point ordinal scale ranges from No symptoms (0) to Death (6), with higher scores representing worse outcome.
Time Frame: 8 Days post subarachnoid hemorrhage (SAH) event
Population: as for outcome 1
Arm/Group | N-acetylcysteine IV Infusion at 0.5 gm Hourly | Placebo for N-acetylcysteine IV Infusion at 0.5 gm Hourly | Acetaminophen Plus N-acetylcysteine IV Infusion
Number analyzed (Participants) | 0 | 0 | 0

5. Primary Outcome: Glasgow Outcome Scale (GOS) Score
Description: The Glasgow Outcome Scale (GOS) is a scale used to assess recovery of participants with brain damage. The scale has 5 categories: Death (1), Persistent vegetative state (2), Severe disability (3), Moderate disability (4), Good recovery (5).
Time Frame: 8 Days post subarachnoid hemorrhage (SAH) event
Population: as for outcome 1
Arm/Group | N-acetylcysteine IV Infusion at 0.5 gm Hourly | Placebo for N-acetylcysteine IV Infusion at 0.5 gm Hourly | Acetaminophen Plus N-acetylcysteine IV Infusion
Number analyzed (Participants) | 0 | 0 | 0

6. Primary Outcome: The Barthel Index Score
Description: The Barthel index measures the extent to which someone can function independently during basic activities of daily living. Scores range from (from 0 to 100), 0 meaning disability and 100 meaning independence, therefore, higher score, better outcome.
Time Frame: 8 Days post subarachnoid hemorrhage (SAH) event
Population: as for outcome 1
Arm/Group | N-acetylcysteine IV Infusion at 0.5 gm Hourly | Placebo for N-acetylcysteine IV Infusion at 0.5 gm Hourly | Acetaminophen Plus N-acetylcysteine IV Infusion
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline to 21 days
Description: Adverse event information was collected for any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research. Adverse events were collected from the time the consent was signed through participant completion.
Arm/Group | N-acetylcysteine IV Infusion at 0.5 gm Hourly | Placebo for N-acetylcysteine IV Infusion at 0.5 gm Hourly | Acetaminophen Plus N-acetylcysteine IV Infusion
All-Cause Mortality (participants affected / at risk) | 3/16 | 6/17 | 0/11
Serious Adverse Events (participants affected / at risk) | 1/16 | 4/17 | 2/11
Other Adverse Events (participants affected / at risk) | 1/16 | 1/17 | 1/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | N-acetylcysteine IV Infusion at 0.5 gm Hourly (N=16) | Placebo for N-acetylcysteine IV Infusion at 0.5 gm Hourly (N=17) | Acetaminophen Plus N-acetylcysteine IV Infusion (N=11)
Vasospasm (Nervous system disorders) | 0 | 2 | 1 — Subarachnoid hemorrhage related vasospasm putting the patient at risk of stroke
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Death (General disorders) | 1 | 2 | 0
Ischemic Stroke (Nervous system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | N-acetylcysteine IV Infusion at 0.5 gm Hourly (N=16) | Placebo for N-acetylcysteine IV Infusion at 0.5 gm Hourly (N=17) | Acetaminophen Plus N-acetylcysteine IV Infusion (N=11)
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
The original trial had multiple stops and starts in enrollment due to PI relocation and funding gaps. This prolonged the patient enrollment periods. Further, the original PI unexpectedly passed away quite suddenly at which point the data management and supervision of the trial reporting passed to its current reporting physician.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-29): https://cdn.clinicaltrials.gov/large-docs/59/NCT00585559/Prot_SAP_000.pdf